CLINICAL TRIAL: NCT05670834
Title: Association Between Matrix Metalloproteinase-2 Gene Polymorphism rs243865 and Susceptibility to Cataract Development
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Tasneem Sayed Hawwary Ahmed, demonstrator, Sohag University
Other Study IDs: Soh-Med-22-12-06
Record Dates: First submitted 2022-12-15; First posted 2023-01-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample will be obtained from all participants by withdrawing 3 mL of blood via venipuncture in EDTA tube
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group (GroupA): normal healthy non-cataractous volunteers aged ≥21 years
  Interventions: Genetic: genotyping assay by real-time PCR; Diagnostic Test: ELISA
- Group B (experimental group 1): cataractous patients aged >50 years and diagnosed with senile cataract.
  Interventions: Genetic: genotyping assay by real-time PCR; Diagnostic Test: ELISA
- Group C (experimental group 2): cataractous patients aged ≥21 to 50 years and diagnosed with secondary cataract
  Interventions: Genetic: genotyping assay by real-time PCR; Diagnostic Test: ELISA

INTERVENTIONS:
Genetic: genotyping assay by real-time PCR — genotyping assay of MMP-2 gene with the real-time polymerase chain reaction
Diagnostic Test: ELISA — . IL-6 level in serum will be analyzed by ELISA assay kit.

SUMMARY:
The primary aim of this study is to investigate the potential association between MMP-2 gene polymorphism and susceptibility to cataract development in Egyptian patients. Furthermore, this study aims to compare between cataract patients and healthy controls by measuring the serum IL-6 concentration to evaluate its relationship with disease.

DETAILED DESCRIPTION:
Cataract is a leading cause of blindness worldwide and is more common in low socioeconomic states and developing countries. According to the WHO, among 3 million visually impaired and 1 million blind persons in Egypt, about 60% have cataract.

The lens undergoes several morphological, biochemical, and physical changes with age which are causal for the formation of age-related cataract.

Oxidative stress can directly influence the solubility of the lens proteins, which increases the lens's opacity.

some studies suggest that inflammatory response may be involved in the occurrence of catarac. and that the pathophysiology is largely attributed to peptide mediators, such as transforming growth factor-beta (TGF-β), epidermal growth factor (EGF) and matrix metalloproteinases (MMPs), with the inhibition of these and other related molecules showing promising results.

Matrix metalloproteinases (MMPs) are a kind of calcium-zinc ion-dependent proteolytic enzyme involved in a variety of cellular processes. MMPs are well known for their ability to degrade the extracellular matrix (ECM) and are involved in several intracellular mechanisms from cell differentiation, proliferation, and angiogenesis to apoptosis.

Several studies' results suggest that the rs243865 (16q13-q21) polymorphism in the promoter region of the metalloproteinase-2 (MMP-2) gene is associated with ophthalmological disorders such as age-related macular degeneration. A recent study suggested that the MMP-2 rs243865 (C/T) polymorphism is associated with an increased risk of cataract.

The expression and activation of MMP-2 can be regulated by environmental influences from surrounding stroma, such as cytokines. some studies suggest that IL6 upregulates the expression of MMPs including MMP-2.

IL-6 is a soluble mediator with a pleiotropic effect on inflammation, immune response, and hematopoiesis. high levels of Il-6 in cataract patients may support the inflammatory response theory of disease development.

this study will follow the tenets of the Declaration of Helsinki. All study participants will sign informed written consent before enrolment in this study.

All study participants will be subjected to complete ophthalmic examination including slit-lamp and fundus examinations. Detailed medical history will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Group A (control group) will include 30 eyes of 30 normal healthy non-cataractous volunteers aged ≥21 years. Group B (experimental group 1) will include 30 eyes of 30 cataractous patients aged >50 years and diagnosed with senile cataract. Group C (experimental group 2) will include 30 eyes of 30 cataractous patients aged ≥21 to 50 years and diagnosed with secondary cataract. The control group will include participants who will be age-matched and sex-matched with the patients in the experimental groups

Exclusion Criteria:

* concomitant eye pathology or inflammation, systemic diseases and previous eye or systemic surgery.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cataractous patients in Department of ophthalmology in Sohag University Hospitals and healthy controls of matched age and sex
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
MMP-2 gene (rs243865) polymorphism in cataract patients and healthy controls | 1 year maximum
  Matrix Metalloproteinase-2 Gene Polymorphism using real-time PCR

SECONDARY OUTCOMES:
compare between cataract patients and healthy controls by measuring the serum IL-6 concentration to evaluate its relationship with disease. | 1 year maximum
  measure serum levels of IL-6 by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong Y, Mu GY, Chen F, Zhao RL, Wang M, Wang B. Correlation between MMP-2 gene polymorphism and cataract susceptibility. Eur Rev Med Pharmacol Sci. 2019 Apr;23(8):3167-3172. doi: 10.26355/eurrev_201904_17674. PMID 31081067